CLINICAL TRIAL: NCT06717958
Title: A Prospective, Single-arm, Open-label, Multicenter Phase II Trial Evaluating the Efficacy and Safety of Ivosidenib Maintenance Therapy After Allogeneic Stem Cell Transplantation (alloSCT) in Patients With Acute Myeloid Leukemia (AML) and Myelodysplastic Neoplasia (MD) Carrying an IDH1 Mutation
Brief Title: Prospective Evaluation of Ivosidenib Maintenance Following Allogeneic Stem Cell Transplantation in Patients With Acute Myeloid Leukemia or High-risk Myelodysplastic Neoplasia With IDH1 (Isocitrate Dehydrogenase 1) Mutation
Acronym: PIVOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-PIVOT1-085
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: AML; MDS
MeSH Terms: interventions — ivosidenib; Magnesium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivosidenib (Experimental)
  Interventions: Drug: Ivosidenib 250 MG (milligram)

INTERVENTIONS:
Drug: Ivosidenib 250 MG (milligram) — oral

SUMMARY:
maintenance of AML or MDS patients with known IDH1 mutation after allogeneic stem cell transplantation within past 100 days

DETAILED DESCRIPTION:
Determination of the efficacy of Ivosidenib to improve event-free survival when given as maintenance therapy following alloSCT.

ELIGIBILITY:
Inclusion criterion:

* AML or MDS with IDH1 mutation

Exclusion criteria:

* active GvHD (graft vs host disease) grade III-IV according to Harris criteria requiring steroids >1mg/ kg prednisolone equivalent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
event-free survival | 24 months

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (12):
  - Universitätsklinikum Aachen, Aachen
  - Technische Universitaet Dresden, Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Essen, Essen
  - Martin-Luther-Universitaet Halle-Wittenberg, Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universität Leipzig, Leipzig
  - Klinikum der Technischen Universitaet Muenchen (TUM Klinikum), München
  - Universität Münster, Münster
  - Rostock University Medical Center, Rostock
  - Universitaetsklinikum Ulm, Ulm